CLINICAL TRIAL: NCT01627210
Title: Evaluation of Glycemic Control Using Adjunctive Continuous Glucose Monitoring With the Dexcom G4 System - GLYCOAIM Study
Brief Title: Evaluation of Glycemic Control Using Adjunctive Continuous Glucose Monitoring With the Dexcom G4 System
Acronym: GLYCOAIM
Status: Completed | Type: Observational
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL900920
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, non-randomized, observational study conducted in the United States.Up to sixty (60) subjects will be enrolled. The purpose of the study is to evaluate long-term utility and usability of Dexcom G4 Continuous Glucose Monitoring (CGM) System. Subjects will be followed monthly over a period of one year.

ELIGIBILITY:
Inclusion Criteria:

* Require intensive insulin therapy, defined as use of Continuous Subcutaneous Insulin Infusion (CSII) i.e. insulin pumps or multiple daily injections (MDI.
* Willing to refrain from use of any acetaminophen - containing (ACT) medication during the study, up to 24-hours before the initial sensor insertion.

Exclusion Criteria:

* Have extensive skin changes/ diseases that preclude wearing the device.
* Dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the Dexcom G4 system utility and usability during home use. | One year
  The primary object of the study is to evaluate the Dexcom G4 system utility and usability during home use. Variables to be evaluated are sensor used, length of use, and data capture during use.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Catalina Research Institute, Chino, California
  - Diabetes and Endocrine Associate, La Mesa, California
  - Infosphere, West Hills, California
  - Desert Endocrinology Clinical Research Center, Henderson, Nevada